CLINICAL TRIAL: NCT03756766
Title: REspiratory Syncytial Virus Consortium in EUrope (RESCEU):Presumed Risk Factors and Biomarkers for RSV-related Severe Disease and Related Sequelae
Brief Title: Understanding RSV: Severe Disease and the Long Term Consequences
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Innovative Medicines Initiative (Other); Respiratory syncytial virus consortium in Europe (Unknown)
Responsible Party: Sponsor
Other Study IDs: OVG 2017/02
Record Dates: First submitted 2018-10-04; First posted 2018-11-28 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-01

CONDITIONS: Respiratory Syncytial Virus (RSV)
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants that enrol in Group 1 will have additional consent to retain specimens for the biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RSV positive ARTI: RSV point of care testing will be performed (if result not already available) to confirm RSV positive status. Individuals with confirmed acute respiratory tract infection (ARTI) secondary to RSV (Group 1- active) will have nasopharyngeal swabs, blood samples, urine samples and stool samples taken at the time of recruitment and again at 7 weeks (convalescence).
  Group 1 participants are categorised into 4 groups as follows:
  Group 1a and 1b participants are healthy infants with an RSV infection either requiring hospitalisation for at least 12 hours or not requiring hospitalisation respectively.
  Group 1c & 1d are infants with an RSV infection with any co-morbidity that would exclude them from Group 1a and 1b either requiring hospitalisation for at least 12 hours or not respectively.
  Interventions: Diagnostic Test: RSV point of care testing
- Healthy controls: This group will include healthy infants (Group 2) who do not have an RSV positive respiratory tract infection and have been asymptomatic in the week preceding and following recruitment.
  This group will have nasopharyngeal swabs, a blood test and a stool and urine sample taken at enrolment only.

INTERVENTIONS:
Diagnostic Test: RSV point of care testing — Patients will have 2 nasopharyngeal swabs, a nasal swab, a stool and urine taken at baseline/ enrolment and the RSV positive ARTI group will have samples repeated at 6-8weeks.
  Other Names: Venepuncture; Nasopharyngeal swabs; stool sample; Urine sample
  Groups: RSV positive ARTI

SUMMARY:
The study design is a case-control, sample based study. 275 cases (Group 1), infants <12 months old with RSV infection and 40 controls (Group 2), otherwise healthy infants <12 months old without RSV infection will be recruited. Samples will be taken on enrolment and for infants in Group 1; repeated at 7 weeks convalescence. There will be annual follow up by questionnaire for up to 6 years and a minimum of 1 year, depending at what stage in the study the infant is enrolled.

DETAILED DESCRIPTION:
Human respiratory syncytial virus (RSV) causes severe disease in the very young, elderly and in high risk groups. Worldwide in 2005 there were an estimated 34 million cases of acute lower respiratory tract infection (ALRI), 3.4 million ALRI hospitalisations and 55,000 to 199,000 deaths associated with RSV in children <5 years old. RSV infection in childhood is associated with subsequent wheezing and asthma. These long-term sequelae pose a substantial additional burden on healthcare systems. There is a parallel need to assemble clinical resources to identify the correlates of severe RSV disease for clinical management, classification of disease severity in clinical trials and identification of biomarkers for severe disease, which are currently lacking.

Group 1: Infants under 12 months with an RSV infection will have nasopharyngeal swabs, blood, urine and stool samples taken at the onset of infection and again 6 - 8 weeks later, in convalescence. An online diary will be completed for 2 weeks during illness to record the participant and parent health. The participant and their family will be followed up annually by questionnaire, for a maximum of 6 years. When the study data are analysed, the infants will be subdivided into 4 further groups; healthy infants requiring hospitalisation, healthy infants not requiring hospitalisation, infants with co-morbidity, requiring hospitalisation and infants with a co-morbidity not requiring hospitalisation. Group 2: Well, healthy infants, under 12 months with no acute respiratory infection will have nasopharyngeal swab,blood, urine and stool samples taken on enrolment. They will receive a follow up contact 7 days after enrolment to assess if they have developed any illness. The participant and their family will be followed up annually by questionnaire, for a maximum of 6 years.

ELIGIBILITY:
Inclusion Criteria: All of the following must apply

* parent/carer of the infant is willing and able to give informed consent for participation in the study
* Male or female, less than 12 months of age at enrolment
* Parent has a telephone

For group 1 only:

* Hospitalised for <48 hours at enrolment or within 96 hours of onset of illness
* Live near enough to a participating study centre for the 6-8 week home visit

Exclusion Criteria:

* Infants who have received treatment for RSV infection (eg: ribavirin)
* Infants who have had prior exposure to an RSV vaccine or medication
* Infants who have received preventative therapy for RSV (eg; palivizumab)
* Infants who have received oral steroids or montelukast within 7days of enrolment on the study

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants less than 12 months old who present to their GP of to hospital with RSV positive respiratory disease.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Estimated)
Dates: Start 2017-12-19 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Ribonucleic acid (RNA) transcripts (Transcriptomics) that are up and down regulated in severe RSV infection | 8 weeks
  Analysis of blood to determine cellular expression of RNA during a severe, acute RSV respiratory tract infection
Cellular protein concentration changes (proteomics) in response to severe RSV infection | 8 weeks
  Analysis of blood samples to determine how cellular protein concentrations change in response to severe RSV infection
Cellular metabolite concentration changes associated with severe RSV disease | 8 weeks
  Analysis of urine and blood to identify which metabolic pathways are up-regulated at a cellular level following severe RSV infection. This is determined by measuring metabolic by-products
The relationship between infant RSV infection of different severity and school age asthma | Year 6
  Symptoms of asthma, diagnosis and use of asthma medication will be measured by parental questionnaire/medical records.

SECONDARY OUTCOMES:
Ribonucleic acid (RNA) transcripts that are up or down regulated and contribute to respiratory sequelae following RSV infection in infants | 3 years
  Analysis of blood samples will determine changes in cellular RNA associated with RSV infection.
Cellular protein concentration changes (Proteomics) affecting respiratory sequelae following RSV infection in infants | 3 years
  Analysis of blood to determine how cellular protein production is up or down regulated in response to RSV infection to correlate with subsequent respiratory sequelae
Cellular metabolite concentration changes that contribute to respiratory sequelae following RSV infection | 3 years
  Analysis of blood and urine to determine which cellular metabolites are produced in increasing quantities during RSV infection and which are subsequently responsible for respiratory sequelae.
Respiratory sequelae following RSV infection in infants | 3 years
  Respiratory sequelae in participants will be determined by completion of a baseline questionnaire followed by an annual questionnaire for a maximum of 3 years.
  The questionnaires record patient demographics, number of siblings, family history of atopy, exposure to household smoke and pets and the ability of the child and family members to complete their usual activities
Viral load associated with mild and severe RSV disease | 8 weeks
  Nasopharyngeal swabs will be taken at baseline and at 6-8weeks to measure viral load
Genetic sequence of RSV associated with mild and severe disease | 8 weeks
  Nasopharyngeal samples will be taken at baseline and at 6-8weeks do determine the genetic sequencing of the Respiratory Syncytial Virus.
Cellular immune response during RSV infection | 8 weeks
  Whole blood will be used for flow cytometric cell phenotyping to determine which immune cells are activated in response to RSV
Cytokine release associated with severe RSV disease | 8 weeks
  Whole blood will be used to perform intracellular cytokine staining in response to RSV infection
Altered gene expression associated with severe RSV disease | 8 weeks
  Blood sampling to determine epigenetic changes associated with RSV infection
RSV disease severity | 8 weeks
  This is determined using a standardized respiratory clinical severity score (ReSVinet) which is performed at baseline.
  This score has 7 subscales;
  1. Feeding intolerance (Score 0-3)
  2. Medical intervention (score 0-3)
  3. Respiratory difficulty (score 0-3)
  4. Respiratory frequency (score 0-3)
  5. Presence of apnoea (either 0, or 3)
  6. General condition (score 0-3)
  7. fever (0-2) The total score is determined by adding each component part. The total score is from 0-20. A score of 0 reflects very mild disease whilst a score of 20 indicates severe disease
Health care costs and resource use | 3 years
  This will be determined using annual questionnaires sent to participants. The questions include: visits to healthcare providers (hospital, GP), number of admissions and duration where applicable and medication use.
Interruption to normal activities associated with RSV disease | 3 years
  Baseline parental questionnaire followed by 14 day symptom diary at onset of illness. Subsequent annual questionnaire for total of 3 years to determine subsequent disease sequelae.
  These questionnaires record symptom severity, duration of symptoms, whether the symptoms affect activities of daily living and a record of persisting symptoms. The follow up questionnaires will extract information about subsequent respiratory symptoms (cough, wheeze), whether the participant has required subsequent review by a healthcare practitioner or been admitted to hospital and during of admission. It also records the need for ongoing medications.
  The information extracted is qualitative in nature. There is no scale used for recording this information.
Compare the incidence of asthma after RSV hospitalisation with incidence of asthma following hospitalisation for viral infections | Year 4
  Parental questionnaires and participant medical records
Compare the incidence of asthma after RSV hospitalisation with incidence of asthma following hospitalisation for viral infections | Year 5
  Parental questionnaires and participant medical records
Compare the incidence of asthma after RSV hospitalisation with incidence of asthma following hospitalisation for viral infections | Year 6
  Parental questionnaires and participant medical records
Risk factors for persistent wheeze at 3 and 6 years of age | Year 4
  Demographic and clinical parameters and outcomes from CRF/demographic questionnaires
Risk factors for persistent wheeze at 3 and 6 years of age | Year 5
  Demographic and clinical parameters and outcomes from CRF/demographic questionnaires
Risk factors for persistent wheeze at 3 and 6 years of age | Year 6
  Demographic and clinical parameters and outcomes from CRF/demographic questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pollard, Study Chair — Oxford Vaccine Group
Locations (2):
- United Kingdom (2):
  - Oxford University Hospitals NHS Trust, Oxford
  - Oxford Vaccine Group, Centre for Clinical Vaccinology and Tropical Medicine, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data sets will be shared with other researchers within the RESCEU consortium. These data sets will include information from participants baseline and annual questionnaires and results from bloods, respiratory samples, urine and stool specimens taken at onset of RSV illness and at 6-8 weeks convalescence.
Supporting Information: Study Protocol
Time Frame: Data will be shared between researchers within the RESCEU consortium as soon as available during the study period. This is currently ongoing. Sharing of the final study information will occur 12-24 months after completion.
Access Criteria: During the study period only researchers involved within the RESCEU consortium will have access to the anonymised individual participant data.

REFERENCES:
- [Derived] McGinley JP, Lin GL, Oner D, Golubchik T, O'Connor D, Snape MD, Gruselle O, Langedijk AC, Wildenbeest J, Openshaw P, Nair H, Aerssens J, Bont L, Martinon-Torres F, Drysdale SB, Pollard AJ; RESCEU Investigators. Clinical and Viral Factors Associated With Disease Severity and Subsequent Wheezing in Infants With Respiratory Syncytial Virus Infection. J Infect Dis. 2022 Aug 12;226(Suppl 1):S45-S54. doi: 10.1093/infdis/jiac163. PMID 35902389
- [Derived] Jefferies K, Drysdale SB, Robinson H, Clutterbuck EA, Blackwell L, McGinley J, Lin GL, Galal U, Nair H, Aerssens J, Oner D, Langedijk A, Bont L, Wildenbeest JG, Martinon-Torres F, Rodriguez-Tenreiro Sanchez C, Nadel S, Openshaw P, Thwaites R, Widjojoatmodjo M, Zhang L, Nguyen TL, Giaquinto C, Giordano G, Baraldi E, Pollard AJ; RESCEU Investigators. Presumed Risk Factors and Biomarkers for Severe Respiratory Syncytial Virus Disease and Related Sequelae: Protocol for an Observational Multicenter, Case-Control Study From the Respiratory Syncytial Virus Consortium in Europe (RESCEU). J Infect Dis. 2020 Oct 7;222(Suppl 7):S658-S665. doi: 10.1093/infdis/jiaa239. PMID 32794560
- [Derived] Lin GL, Golubchik T, Drysdale S, O'Connor D, Jefferies K, Brown A, de Cesare M, Bonsall D, Ansari MA, Aerssens J, Bont L, Openshaw P, Martinon-Torres F, Bowden R, Pollard AJ; RESCEU Investigators. Simultaneous Viral Whole-Genome Sequencing and Differential Expression Profiling in Respiratory Syncytial Virus Infection of Infants. J Infect Dis. 2020 Oct 7;222(Suppl 7):S666-S671. doi: 10.1093/infdis/jiaa448. PMID 32702120
- See also: RESCEU website (coordinators of the Understanding RSV study) — http://resc-eu.org/